CLINICAL TRIAL: NCT07086963
Title: Is Dorsal Inlay Graft (DIG) With TIP Repair Superior to TIP Alone for Primary Hypospadias? A Randomized Clinical Trial
Brief Title: Is Dorsal Inlay Graft (DIG) With TIP Repair Superior to TIP Alone for Primary Hypospadias?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammad Daboos (Other)
Responsible Party: Sponsor-Investigator, Mohammad Daboos, Assistant professor of pediatric surgery, Pediatric Surgery Department, Al-Azhar University., Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SVU/SUR011/4/22/12/519
Record Dates: First submitted 2025-07-05; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Hypospadias
Keywords: Grafted TIP; Tabularized Incised Plate
MeSH Terms: conditions — Hypospadias | interventions — Lysine Acetyltransferase 5

STUDY DESIGN:
Intervention Model Description: Group 1: Repaired with standard TIP repair as described by Snodgrass Group 2: Repaired with TIP with GIP using preputial graft
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Repaired with standard Tubularized incised plate repair as described by Snodgrass
  Interventions: Procedure: Repaired with standard TIP repair as described by Snodgrass
- Group 2 (Active Comparator): Repaired with Grafted Tubularized incised plate repair using preputial graft
  Interventions: Procedure: Repaired with TIP with GIP using preputial graft

INTERVENTIONS:
Procedure: Repaired with standard TIP repair as described by Snodgrass — Urethroplasty was performed over a 6-8 Fr Nelaton catheter (according to patient age and glans size) using 7/0 subcuticular continuous suture. Adequate meatus was left around the urethral catheter at the glans tip, followed by spongioplasty and a second-layer dartos fascia coverage.
  Mucosal collar approximation and skin closure Glanular closure was then initiated with deep but superficial stitches using 7/0 or 6/0 polyglactin suture, and mucosal suture closure. Skin closure was achieved by preparing viable skin while avoiding midline skin closure by preparing a vascularized preputial skin flap to avoid skin coverage complications with subsequent UCF
  Arms: Group 1
Procedure: Repaired with TIP with GIP using preputial graft — The urethral plate was deeply incised from the glans tip, extending downwards beyond the junction between the plate and the hypospadiac meatus Graft fixation The graft was then spread to cover the raw area and fixed to the edges of the urethral plate.
  Urethroplasty was performed over a 6-8 Fr Nelaton catheter (according to patient age and glans size) using 7/0 subcuticular continuous suture. Adequate meatus was left around the urethral catheter at the glans tip, followed by spongioplasty and a second-layer dartos fascia coverage.
  Mucosal collar approximation and skin closure Glanular closure was then initiated with deep but superficial stitches using 7/0 or 6/0 polyglactin suture, and mucosal suture closure. Skin closure was achieved by preparing viable skin while avoiding midline skin closure by preparing a vascularized preputial skin flap to avoid skin coverage complications with subsequent UCF
  Arms: Group 2

SUMMARY:
This prospective, randomized study included all patients who presented with primary hypospadias without chordee, Patients were randomized into two groups as group 1 or group 2,Group 1: Repaired with standard TIP repair as described by Snodgrass Group 2: Repaired with TIP with GIP using preputial graft. In both groups the functional outcomes were primarily compared regarding meatal position, shape, and the functional outcomes of the neourethra, in addition to other complications such as UCF, wound complications, cosmetic results and the need for a second surgery.

the investigators aimed to investigate whether GIP with TIP repair is superior to TIP, as described by Snodgrass in different types of UP and to provide an overview of the technical aspects of current TIP repair practices.

DETAILED DESCRIPTION:
This prospective, randomized study included all patients who presented with primary hypospadias without chordee.

investigators aimed to investigate whether grafted inlay patch with Tabularized Incised Plate repair is superior to TIP, as described by Snodgrass in different types of UP and to provide an overview of the technical aspects of current TIP repair practices.

Patients were randomized into two groups as group 1 or group 2,Group 1: Repaired with standard TIP repair as described by Snodgrass Group 2: Repaired with TIP with GIP using preputial graft. Patients were randomized into two groups using sealed envelopes labeled as group 1 or group 2, selected by the operating theater chief nurse. An independent statistician approved the sample size.

In both groups the functional outcomes were primarily compared regarding meatal position, shape, and the functional outcomes of the neourethra, in addition to other complications such as UCF, wound complications, cosmetic results and the need for a second surgery.

The first visit occurred on the 5th postoperative day. On 2nd week, the patients attended for catheter removal after complete healing. Calibration was performed one week after catheter removal, followed by monthly for the first six months, with HOSE scoring conducted after six months.

ELIGIBILITY:
Inclusion Criteria:

* Primary hypospadias candidates for one-stage repair
* Uncircumcised cases
* Pediatric age group
* Patients with regular follow up

Exclusion Criteria:

* The presence of chordee or urethral anomalies requiring division of the urethral plate or staged repair
* Small glans < 11mm
* glanular hypospadias

Ages: 6 Months to 120 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 584 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2025-07-25 (Estimated); Study Completion 2025-08-08 (Estimated)

PRIMARY OUTCOMES:
Surgical outcomes | 6 months
  complications rates
cosmetic results | 6 months
  cosmetic results with Hypospadias Objective Scoring Evaluation.
Functional outcomes | 6 months
  Urine Flow from the neourethra

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Daboos, Principal Investigator — Al-Azhar University
Locations (1):
- Mohammad Daboos, Cairo, Egypt

REFERENCES:
- [Derived] Negm MA, Abdelrasheed AA, Daboos M, Khedre MM, Abdelrahman MF, Abo-Halawa NAE, Ibrahim IA, Shehata MA. Is dorsal inlay graft (DIG) with TIP repair superior to TIP alone for primary hypospadias? A randomized clinical trial. BMC Pediatr. 2026 Jan 26. doi: 10.1186/s12887-025-06247-7. Online ahead of print. PMID 41588344